CLINICAL TRIAL: NCT05012046
Title: Effect of 100% Orange Juice Intake on Subjective Appetite, Food Intake, Glycemic Response and Subjective Mood in Healthy Adults
Brief Title: Effect of 100% Orange Juice on Food Intake and Glycemic Response in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB: 2021-177
Record Dates: First submitted 2021-08-11; First posted 2021-08-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Healthy; Adult; Glycemic Response; Appetite
Keywords: Food intake; Appetite; Blood glucose; Glycemic response; Orange juice; Adults
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orange juice (Experimental): Treatment beverage
  Interventions: Other: Orange juice
- Orange flavoured drink (Experimental): Treatment beverage
  Interventions: Other: Orange flavoured drink
- Water (Experimental): Treatment beverage
  Interventions: Other: Water

INTERVENTIONS:
Other: Orange juice — Matched for volume (240 mL/ 8 oz) of other test beverages. 100% orange juice.
  Arms: Orange juice
Other: Orange flavoured drink — Matched for volume (240 mL/ 8 oz) of other test beverages. Orange flavoured drink
  Arms: Orange flavoured drink
Other: Water — Matched for volume (240 mL/ 8 oz) of other test beverages. Water control
  Arms: Water

SUMMARY:
The purpose of this study is to determine the effects of 100% orange juice on short-term food intake (FI), satiety, post-prandial glycemia and mood in healthy adults. We hypothesize that the consumption of 100% orange juice in the pre-meal environment will improve satiety signals and mood, and suppress FI through its effect on post-prandial glycemia.

DETAILED DESCRIPTION:
A randomized within-subjects repeated measures design will be employed. Study visits will take place in the morning, separated one-week apart. At each session, participants will consume one of three treatments: 1) 100% orange juice; 2) orange flavoured drink; or 3) water. Glycemic response will be measured for 60 minutes (baseline (0 minutes), 15 minutes, 30 minutes, 45 minutes and 60 minutes) post-treatment via finger prick. Blood glucose measures will also be provided over 24 hours via a Dexcom G6 continuous glucose monitoring (CGM) device. Subjective appetite, emotions and mood will be measured for 90 minutes min (baseline (0 minutes), 15 minutes, 30 minutes, 45 minutes, 60 minutes and 90 minutes) post-treatment. At 60 minutes, participants will consume an ad libitum pizza lunch to evaluate food intake. After lunch, participants will be sent home with a rest-of-the-day food intake sheet to record their snacks, meals, and beverages, as well as a physical activity log to record their physical activity for the rest of the day following test session completion.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years;
* within the healthy body mass index (BMI) range for adults of 18.5-24.9 kg/m2.

Exclusion Criteria:

* individuals who are dieting;
* restrained eaters;
* breakfast skippers;
* those who dislike breakfast or lunch treatment foods;
* those taking medication;
* individuals with any metabolic disorders or significant weight fluctuations.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline glycemic response (acute phase) | Collected at baseline (0 minutes), 15 minutes, 30 minutes, 45 minutes, and 60 minutes post-treatment consumption
  Blood glucose (mmol/L). Three drops of blood from the finger will be collected at each time point using a single-use, auto-disabling lancet device and sodium fluoride/potassium oxalate capillary blood collection tubes. Blood glucose will be measured using a YSI 2900D Biochemistry Analyzer (YSI Inc., Yellow Springs, OH).
Rest-of-day blood glucose concentrations | Continuous measurements for 24 hours post-treatment consumption
  Blood glucose (mmol/L). Rest-of-day blood glucose concentrations will be determined using a Dexcom G6 CGM system.
Ad libitum food intake | At 60 minutes post-treatment consumption
  Lunch pizza meal. Food intake will be determined by weighing the meal before and after serving. The net weight of the test meal will be converted to calories.

SECONDARY OUTCOMES:
Change from baseline subjective appetite | Collected at baseline (0 minutes), 15 minutes, 30 minutes, 45 minutes, and 60 minutes post-treatment consumption
  Measured using visual analogue scales (VAS). Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings. Questions will include desire to eat, fullness, hunger, and prospective food consumption. Individual questions will be used to form a composite score.
Change from baseline subjective emotions and mood | Collected at baseline (0 minutes), 15 minutes, 30 minutes, 45 minutes, and 60 minutes post-treatment consumption
  Measured using visual analogue scales. Each VAS is a 100 mm line where they will place a pencil mark to describe their feelings. Questions will measure aggression, anger, excitement, disappointment, frustration, alertness, sadness, tension, effort, happiness, weariness, calmness, sleepiness, and wellness. Individual questions will be used to form a composite score.
Rest-of-the-day food intake | For the rest of the day following test session completion (1 day)
  Participants will be sent home with a rest-of-the-day food intake recall sheet to record their snacks, meals, and beverages.
  Rest of day food log
Rest-of-the-day physical activity | For the rest of the day following test session completion (1 day)
  Participants will be sent home with a rest-of-the-day physical activity recall sheet to record any activities performed.
  Physical activity questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Centre for Urban Innovation (CUI-109), School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No